CLINICAL TRIAL: NCT05417048
Title: miRNAs of Circulating Glycosylated Extracellular Vesicles as Biomarkers for Early Diagnosis of Breast Cancer Patients
Brief Title: Clinical Study of Glycosylated Extracellular Vesicles for Early Diagnosis of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Beijing Glyexo Gene Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Tao OUYANG, Director of Breast Center of Peking University Cancer Hospital, Peking University
Other Study IDs: BC-P31
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of blood of patients before treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breat cancer: Histologically confirmed breast cancer patients(Stage I-III)
  Interventions: Diagnostic Test: Blood Sample
- Benign breast disease: Histologically confirmed breast fibroma, intraductal papilloma,mammary hyperplasia, breast cyst etc
  Interventions: Diagnostic Test: Blood Sample
- Healthy control: No breast lesions detected by clinical examination/mammography/ultrasound/breast magnetic resonance imaging (MRI)
  Interventions: Diagnostic Test: Blood Sample

INTERVENTIONS:
Diagnostic Test: Blood Sample — Up to 5mL of blood via venipuncture

SUMMARY:
This is a prospective, single-center, non-randomized, cohort study designed to evaluate the clinical diagnostic performance of glycosylated extracellular vesicles and their contents for early detection of breast cancer.

DETAILED DESCRIPTION:
Early screening technology can improve the survival rate of breast cancer patients. Traditional mammography and ultrasonography have limitations on performance in clinical practice. Extracellular vesicles, one of the three major resources of liquid biopsy, contain multi-omics information that can be used to discover effective biomarkers for early diagnosis and screening of cancers.

In this study, we are going to isolate glycosylated extracellular vesicles from serum of cancer patients and non-cancer people with the novel GlyExo-Capture technology, and perform miRNA sequencing to selected out breast cancer-related markers. Then an early diagnosis model of breast cancer based on the GlyExo-Capture platform is able to be established using machine learning techniques and validated by qPCR experiments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients≥18 years old；
2. Histologically confirmed breast cancer patients，Benign breast disease （ig. breast fibroma, intraductal papilloma,mammary hyperplasia, breast cyst）or No breast lesions detected by clinical examination/mammography/ultrasound/breast magnetic resonance imaging (MRI)
3. Previous not received preoperative radiotherapy, chemotherapy, endocrine therapy, immunotherapy, or other anticancer treatments.
4. Subjects signed informed consent；

Exclusion Criteria:

1. A history of prior or concomitant malignancies;
2. advanced stage breast cancer (stage IV)；
3. Patients were accompanied by severe organic diseases such as heart and cerebral disease, and liver and kidney disease.；
4. Pregnant or lactating women ；
5. Suspected or confirmed lesion was surgically removed；
6. Patients with incomplete clinical data；
7. Patients with poor compliance；
8. Patients with severe mental illness；
9. Patients had received blood transfusions during one month一；

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breat cancer, Benign breast disease and Healthy control
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance of the blood assay for differentiating benign and malignant breast disease using glycosylated extracellular vesicles analysis | 24 months
  The efficacy of the blood-based assay comparing with patholgic diagnosis, the gold standard, and imaging diagnosis, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoqing Fan, MD, Principal Investigator — Breast center at Peking University Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China